CLINICAL TRIAL: NCT05442151
Title: Evaluation Using FAPI-PET Targeting Cancer-associated Fibroblasts
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tadashi Watabe (Other)
Responsible Party: Sponsor-Investigator, Tadashi Watabe, Assistant Professor, Osaka University
Organization: Osaka University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 21472
Record Dates: First submitted 2022-06-18; First posted 2022-07-01 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Neoplasms
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- FAPI-PET/CT group (Other)
  Interventions: Drug: PET/CT ([F-18]FAPI-74)

INTERVENTIONS:
Drug: PET/CT ([F-18]FAPI-74) — PET/CT using [18F] FAPI-74 injection

SUMMARY:
PET / CT examination using [18F] FAPI-74 is performed on patients diagnosed with malignant tumor, and the pathological condition is determined by comparing with FDG-PET/CT examination of conventional diagnostic imaging.

DETAILED DESCRIPTION:
Cancer stroma accounts for more than 90% of all tumors, and cancer-related fibroblasts (CAFs) play an important role in the growth and progression of cancer. FAP expressed in CAF has been found to be expressed in many cancers, and [68Ga] FAPI-04 and [18F] FAPI-74, which are PET diagnostic agents for FAP ligand FAPI, have been used all over the world. The purpose of this study is to perform PET / CT using [18F] FAPI-74 injection for patients diagnosed with malignant tumors, mainly pancreatic cancer and gastric cancer to evaluate the pathology in detail by comparing with the FDG-PET/CT.

ELIGIBILITY:
Inclusion Criteria:

Patients who meet any of the following conditions.

1. Patients who have been diagnosed with malignant tumors or suspected of having malignant tumors and have CT or FDG-PET examination.
2. Patients who have been diagnosed with malignant tumor and are scheduled to receive or have undergone anticancer treatment such as chemotherapy or radiation therapy.
3. Patients suspected of recurrence by clinical findings or diagnostic imaging such as CT or FDG-PET after treatment of malignant tumor

Exclusion Criteria:

1. Pregnant women or patients who may be pregnant
2. Pediatric patients requiring sedation
3. Those who are judged to be inappropriate as subjects.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2022-05-09 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Comparison of the uptake on FAPI-PET with conventional imaging | Within 2 hours after administration of [F-18]FAPI-74 injection
  Comparison of SUV (standardized uptake value) of primary site and metastatic lesions between FAPI-PET and FDG-PET
Comparison with pathological specimens | Within one month after FAPI-PET
  Comparison of expression level (staining score) in FAP immunostaining and SUV in FAPI-PET (FAP staining is graded by scoring evaluation: high expression (3 points), moderate expression (2 points), mild expression (1 point), and no significant expression (0 point).)
Time course of uptake on FAPI-PET | Approximately 6 months after initial FAPI-PET
  Time course of uptake on FAPI-PET before and after treatment compared with conventional imaging

CONTACTS AND LOCATIONS:
Locations (1):
- Osaka University Hospital, Suita, Osaka, Japan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Naka S, Watabe T, Lindner T, Cardinale J, Kurimoto K, Moore M, Tatsumi M, Mori Y, Shimosegawa E, Valla F Jr, Kato H, Giesel FL. One-pot and one-step automated radio-synthesis of [18F]AlF-FAPI-74 using a multi purpose synthesizer: a proof-of-concept experiment. EJNMMI Radiopharm Chem. 2021 Aug 21;6(1):28. doi: 10.1186/s41181-021-00142-z. PMID 34420105